CLINICAL TRIAL: NCT02717676
Title: Episiotomy for Prevention of Perineal Tears During Labor in Women With High Striae Gravidarum Score
Brief Title: Prediction of Perineal Tears by Striae Gravidarum Score
Acronym: TSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TSS
Record Dates: First submitted 2016-03-13; First posted 2016-03-24 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Normal Labor
MeSH Terms: interventions — Episiotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Episiotomy
  Interventions: Procedure: Episiotomy
- Group B (No Intervention): no episiotomy

INTERVENTIONS:
Procedure: Episiotomy — episiotomy will be done after crowning of the fetal head
  Arms: Group A

SUMMARY:
Previous studies concluded that striae gravidarum assessment appears to predict the occurrence of perineal tears and recommend training the health personnel to calculate the total striae score which can help them decide if episiotomy is to be given or not. Episiotomy definitely seems to be preventive for perineal tears but giving episiotomy for the same is still debatable as episiotomy in itself is associated with morbidity. the hypothesis is episiotomy done in patients with high score will definitely protects against perineal tears. So, the aim of study is to determine whether assessment of striae gravidarum score could predict occurrence of tears during labor or not, and if episiotomy will prevent perineal tears in women with high score.

ELIGIBILITY:
Inclusion criteria:

1. Multipara
2. Singleton pregnancy
3. Full-term (37- 40 weeks)
4. Average size fetus (2500-4000 gm)
5. Cephalic-vertex presentation
6. Spontaneous onset of labor
7. No scarred uterus
8. No medical diseases as hypertension
9. No obstetric complications as obstructed labor
10. Women accepted to participate in the study

Exclusion criteria:

1. Multiple pregnancy
2. Women with Previous cesarean sections
3. Preterm labor
4. Malpresentation
5. Fetal macrosomia
6. Medical diseases as diabetes and hypertension
7. Women refuse to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04-02 (Actual); Study Completion 2018-06-02 (Actual)

PRIMARY OUTCOMES:
Rate of third and forth degree perineal tears | intraoperative

SECONDARY OUTCOMES:
Rate of first and second degree perineal tears | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes